CLINICAL TRIAL: NCT06299072
Title: 18-40 Years to Assess Whole Grain (WG) Awareness, Consumption Levels, and Dietary Habits Around Breakfast
Brief Title: A Cross-sectional Online Survey Among Saudi Arabian Population in the Age Group 18-40 Years to Assess Whole Grain (WG) Awareness, Consumption Levels, and Dietary Habits Around Breakfast
Status: Completed | Type: Observational
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: PEP-2303
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Diet, Healthy
Keywords: whole grain; breakfast; habit; consumer
MeSH Terms: conditions — Habits | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Quantitative questionnaire

SUMMARY:
In this online survey conducted suing the YouGov consumer insights panel, the primary aims of this study are to provide for the first time an estimate of consumer awareness regarding wholegrains; their definitions and knowledge of potential benefits in the Saudi Arabia adult population and the he estimated consumption amongst Saudi consumers.

Secondary Objectives are to assess the breakfast habit, oat consumption & health concerns amongst Saudi consumers; identify socio-demographic and consumer characteristics associated with breakfast consumption, the types of foods consumed at breakfast, and fill gaps in knowledge regarding breakfast eating habits, commonly consumed breakfast foods.

ELIGIBILITY:
Inclusion Criteria:

* Participants in online panel survey
* Age between 18 and 40 years
* Current resident of urban Saudi Arabia in Jeddah, Riyadh, & Dammam

Exclusion Criteria:

N.A.

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Three cities in Saudi Arabia, with representation across regions, gender, age group, and education status.
Sampling Method: Non-Probability Sample
Enrollment: 814 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Consumer awareness regarding wholegrains | Approximately 20 minutes
  Single online panel survey
Consumer definitions of wholegrains | Approximately 20 minutes
  Single online panel survey
Consumer knowledge of potential benefits of wholegrains | Approximately 20 minutes
  Single online panel survey
Wholegrain consumption | Approximately 20 minutes
  Single online panel survey

SECONDARY OUTCOMES:
Breakfast habits | Approximately 20 minutes
  Single online panel survey
Oat consumption | Approximately 20 minutes
  Single online panel survey
Health concerns | Approximately 20 minutes
  Single online panel survey
Socio-demographics associated with breakfast consumption | Approximately 20 minutes
  Single online panel survey
Consumer characteristics associated with breakfast consumption | Approximately 20 minutes
  Single online panel survey
Types of foods consumed at breakfast | Approximately 20 minutes
  Single online panel survey
Fill gaps in knowledge regarding breakfast eating habits | Approximately 20 minutes
  Single online panel survey
Commonly consumed breakfast foods | Approximately 20 minutes
  Single online panel survey

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Al Dhaheri, PhD, Principal Investigator — College of Medicine and Health Sciences, Abu Dhabi - UAE
Locations (1):
- Remote, no facility visits, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No